CLINICAL TRIAL: NCT00975364
Title: Pilot Study to Investigate Relationship Between Common Folate Gene Polymorphisms, Folate Status and Cellular Folate Speciation
Brief Title: Folate Gene Polymorphisms and Cellular Folate Speciation Pilot Study
Acronym: FolGene
Status: Completed | Type: Observational
Sponsor: Quadram Institute Bioscience (Other)
Responsible Party: Sponsor
Other Study IDs: IFR05/2008; 08/H0310/153; 2008IFR01L
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Single Nucleotide Polymorphism
Keywords: Folate; Methylenetetrahydrofolate reductase; Speciation; Nutrient status; Bioavailability; Polymorphism, single nucleotide

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — One-off blood sample collected. DNA extracted for genotyping of folate metabolism-related gene single nucleotide polymorphisms
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- blood sampling: Consented volunteers provide a one-off blood sample

SUMMARY:
This pilot study is designed to investigate differences in folate-related genes (single nucleotide polymorphisms) and their relationship to the species of folate present on red blood cells.

DETAILED DESCRIPTION:
The main questions to be addressed in this pilot study are:

1. what is the type of folate in red blood cells in individuals with different methylterahydrofolate reductase (MTHFR) genotypes
2. what is the relationship between other folate metabolism-related gene single nucleotide polymorphisms and type (species) of folate found in red blood cells
3. what is the relationship between folate and other B vitamin status, genotype and folate species
4. is there a relationship between serum ferritin status and folate metabolism

Whole blood will be taken from apparently healthy male and female volunteers, aged 18-65, which will be used to determine genotype for various folate metabolism-related genes. Furthermore, the type of folate present on the red blood cells will be assessed, and folate, vitamin B12, riboflavin and serum ferritin status determined.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65
* Males and females
* Body Mass Index greater than 19.5 and less than 40
* Smokers and non-smokers

Exclusion Criteria:

* Pregnancy or been pregnant in last 12 months
* Diabetes
* Parallel participation in another research project if total amount of blood from combined studies is greater than 470ml
* Participation in another research project where blood samples were taken within the past 4 months, unless total blood volume does not exceed 470ml
* Any person related to or living with a member of the study team
* Has donated or intends to donate blood within 16 weeks (prior to or after) the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults (male and female) aged 18-65
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-02; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Relationship between MTHFR TT, CT and CC genotype and red cell folate species | July 2010

SECONDARY OUTCOMES:
Relationship between other folate metabolism related genes and red cell folate species | July 2010
Relationship between folate, B12, riboflavin and ferritin status and red cell folate species | December 2010

CONTACTS AND LOCATIONS:
Overall Officials: Paul Finglas, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Institute of Food Research, Norwich, Norfolk, United Kingdom